CLINICAL TRIAL: NCT03275662
Title: Microbiota-targeted Dietary Strategies to Reduce Inflammatory Markers of Americans: High Fiber vs Fermented Food
Brief Title: Fermented and Fiber-rich Food (FeFiFo) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Justin L. Sonnenburg, Associate Professor of Microbiology and Immunology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 36643
Record Dates: First submitted 2017-09-06; First posted 2017-09-07 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Metabolic Syndrome; Microbiome; Immune Function; Inflammation
MeSH Terms: conditions — Metabolic Syndrome; Inflammation | interventions — Dietary Fiber; Fermented Foods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber Group (Experimental): Participants are asked to increase their usual dietary fiber intake by 20 grams/day.
  Interventions: Behavioral: Dietary Fiber
- Fermented Foods Group (Experimental): Participants are asked to consume 6 servings of fermented foods per day.
  Interventions: Behavioral: Fermented Foods

INTERVENTIONS:
Behavioral: Dietary Fiber
  Arms: Fiber Group
Behavioral: Fermented Foods
  Arms: Fermented Foods Group

SUMMARY:
The primary objective is to contrast the degree to which increased consumption of dietary fiber vs. fermented food can decrease inflammation, increase microbiota diversity and can impact microbiota production of short-chain fatty acids (SCFA), potential normalizers of metabolic and immune dysfunction, in obese and non-obese adults.

DETAILED DESCRIPTION:
The gut microbiota is central to human health, and the modern, industrialized gut microbiota has been linked to numerous chronic diseases that are driven by inflammation. It is likely dietary changes in the last half-century consistent with adoption of the Western diet have had an adverse impact on the gut microbiota. A critically important next step in this field of research is to identify how different dietary interventions can potentially restore healthy features of the gut microbiota in alignment with the optimization of human health. Dietary interventions that target the microbiota and reduce inflammation may reverse or prevent chronic diseases including obesity, metabolic syndrome, and inflammatory bowel disease. This study is designed to elicit and contrast inflammatory markers in blood with the amount of increase in microbiota diversity and related metabolic output achievable by two dietary approaches commonly available to the general population. The results could contribute to dietary recommendations for reversing the chronic disease epidemics of Westernization.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older, both genders, all ethnic backgrounds
* Healthy subjects willing and able to provide blood, as well as stool specimens
* Able to provide signed and dated informed consent.

Exclusion Criteria:

* Body Mass Index higher than 40.
* Vital signs outside of acceptable range at Screening Visit, i.e., blood pressure greater than 160/100, oral temperature greater than 100 degrees F, pulse greater than 100.
* Use of any of the following drugs within the last 6 months:

  1. systemic antibiotics, antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral);
  2. oral, intravenous, intramuscular, nasal or inhaled corticosteroids;
  3. cytokines;
  4. methotrexate or immunosuppressive cytotoxic agents;
  5. large doses of commercial probiotics consumed (greater than or equal to 10e8 cfu or organisms per day) - includes tablets, capsules, lozenges, chewing gum or powders in which probiotic is a primary component.
  6. consumption of > 20 g fiber/day and > 7 servings of fermented foods per week.
* Acute disease at the time of enrollment (defer sampling until subject recovers). Acute disease is defined as the presence of a moderate or severe illness with or without fever.
* Chronic, clinically significant (unresolved, requiring on-going medical management or medication) pulmonary, cardiovascular, gastrointestinal, hepatic or renal functional abnormality, as determined by medical history or physical examination.
* History of cancer except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision.
* Unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet.
* Recent history of chronic alcohol consumption defined as more than five 1.5-ounce servings of 80 proof distilled spirits, five 12-ounce servings of beer or five 5-ounce servings of wine per day.
* Positive test for HIV, HBV or HCV.
* Any confirmed or suspected condition/state of immunosuppression or immunodeficiency ( primary or acquired) including HIV infection.
* Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time.
* History of active uncontrolled gastrointestinal disorders or diseases including:

  1. inflammatory bowel disease (IBD) including ulcerative colitis (mild-moderate-severe), Crohn's disease (mild-moderate-severe), or indeterminate colitis;
  2. irritable bowel syndrome (IBS) (moderate-severe);
  3. persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated);
  4. chronic constipation.

Female who is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Immune profile: Cytokine Response Score (CRS) | Baseline and 10 weeks
  Change from baseline in CRS at 10 weeks

SECONDARY OUTCOMES:
Microbiota metabolites: short-chain fatty acids (SCFA) | Baseline and 10 weeks
  Change from baseline in short-chain fatty acids (SCFA) at 10 weeks.
Microbiota composition | Baseline and 10 weeks
  Change from baseline in 16S rRNA enumeration at 10 weeks, determined using Illumina-based sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Justin L Sonnenburg, PhD, Principal Investigator — Stanford University; Christopher D Gardner, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wastyk HC, Fragiadakis GK, Perelman D, Dahan D, Merrill BD, Yu FB, Topf M, Gonzalez CG, Van Treuren W, Han S, Robinson JL, Elias JE, Sonnenburg ED, Gardner CD, Sonnenburg JL. Gut-microbiota-targeted diets modulate human immune status. Cell. 2021 Aug 5;184(16):4137-4153.e14. doi: 10.1016/j.cell.2021.06.019. Epub 2021 Jul 12. PMID 34256014
- See also: Study description and results summary — https://med.stanford.edu/nutrition/research/completed-studies/fefifo.html